CLINICAL TRIAL: NCT04621318
Title: A Randomised, Double-blind, Three-arm, Parallel Group, Single-dose Study to Compare the Pharmacokinetics, Pharmacodynamics, Safety, Tolerability, and Immunogenicity of Denosumab (SB16, EU Sourced Prolia®, and US Sourced Prolia®) in Healthy Male Subjects
Brief Title: Pharmacokinetics, Pharmacodynamics, Safety, Tolerability, and Immunogenicity Study of SB16 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samsung Bioepis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: SB16-1001
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Healthy
MeSH Terms: interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SB16 (Experimental): SB16 (proposed denosumab biosimilar)
  Interventions: Drug: Denosumab
- EU Prolia (Active Comparator): EU sourced Prolia (denosumab)
  Interventions: Drug: Denosumab
- US Prolia (Active Comparator): US sourced Prolia (denosumab)
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Denosumab — 60 mg, single-dose

SUMMARY:
This study is to compare PK, PD, safety, tolerability, and immunogenicity profiles of SB16, EU sourced Prolia, and US sourced Prolia in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male, aged 28-55 years (inclusive) on the day of signing the informed consent.
2. Have a body weight between 60.0-90.0 kg (inclusive) and a BMI between 20.0-29.9 kg/m2 (inclusive).
3. Have 12-lead ECG results without clinically significant abnormal findings confirmed by the Investigator.
4. Have vital sign results without clinically significant abnormal findings confirmed by the Investigator.
5. Have physical examination results without clinically significant abnormal findings confirmed by the Investigator.
6. Male subjects who have not had surgical sterilisation must be willing to abstain from sexual intercourse or willing to use a condom in addition to having their female partner use another form of contraception, such as an intra-uterine device, oral contraceptive, injectable progesterone, sub-dermal implant, or tubal ligation unless their partners are infertile (confirmed with written verifications) during the treatment period.
7. Willing and able to comply with scheduled visits, treatment plan, clinical laboratory tests, and other study procedures including lifestyle considerations.
8. Able to provide written informed consent, which must be obtained prior to any study related procedures being performed.
9. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted.

Exclusion Criteria:

1. Have a history and/or current presence of clinically significant atopic allergy, hypersensitivity, or allergic reactions (either spontaneous or following drug administration), also including known or suspected clinically relevant drug hypersensitivity to denosumab or to any of the excipients.
2. Have a history of and/or current clinically significant gastrointestinal, renal, hepatic, cardiovascular, haematological, pulmonary, neurologic, metabolic, psychiatric disorder, drug or alcohol abuse, or allergic disease excluding mild asymptomatic seasonal allergies.
3. Have a history of bone disease or any medical condition that can affect bone metabolism (including osteoporosis, osteogenesis imperfecta, osteomalacia, hyperparathyroidism, hyperthyroidism, hypothyroidism, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, Paget's disease of the bone, and malabsorption syndrome).
4. Have a history of malignancy (including lymphoma, leukaemia, and skin cancer).
5. Have ONJ or risk factors for ONJ such as invasive dental procedures or active periodontal disease within 180 days prior to Randomisation.
6. Have bone fractures within 180 days prior to Randomisation.
7. Have a history of serious infection (associated with hospitalisation and/or which required intravenous antibiotics) within 180 days prior to Randomisation.
8. Have a clinically significant active infection (bacterial, viral, or fungal) including skin infections within 28 days prior to Randomisation.
9. Have any systemic or local infection, a known risk for developing sepsis.
10. Have known intolerance to calcium or vitamin D supplements.
11. Have previously been exposed to denosumab (Prolia®/Xgeva®) and its biosimilar.
12. Have previously been exposed to a monoclonal antibody or fusion protein within 270 days (other than denosumab) prior to Randomisation and/or there is confirmed evidence or clinical suspicion of immunogenicity from previous exposure to a monoclonal antibody or fusion protein.
13. Have previously been exposed to an immunosuppressive agent or biological agent (any other than a monoclonal antibody or fusion protein) within 120 days prior to Randomisation.
14. Have received live vaccines(s) within 30 days prior to Randomisation or who will require live vaccine(s) during the study period.
15. Have a personal or family history of prolonged QT interval syndrome or Torsade de Pointes, or family history of sudden death.
16. Have any of the following abnormal laboratory test results:

    1. Albumin-adjusted serum calcium levels below the LLN or above the ULN.
    2. Serum creatinine levels above 1.5 × ULN.
    3. Any other laboratory abnormalities assessed as clinically significant by the Investigator.
17. Have a positive test result for HBsAg, HCV antibody, or HIV 1or 2.
18. Have a history of immunodeficiency.
19. Have had surgery within 90 days prior to Randomisation, and/or plan to have an operation (including invasive dental procedure) during the study period.
20. Have a history and/or current presence of an illness (including, but not limited to respiratory symptoms [e.g., difficulty breathing or persistent cough] or low-grade fever) within 14 days prior to Randomisation that is classified as clinically significant by the Investigator.
21. Have smoked more than 10 cigarettes, 2 cigars, or 2 pipes per day within 90 days prior to Screening.
22. Have regular consumption of alcoholic beverages that exceeds 14 units per week.
23. Have a positive urinary drug screening result or alcohol breath test result at Screening or Day -1.
24. Have taken any prescription medicine or over-the-counter medicines (except paracetamol) that might have an effect on the objectives of the study in the opinion of the Investigator, within 30 days or 10 half-lives of the medication (whichever period is longer) prior to Randomisation. This includes medications such as, but not limited to: Bisphosphonates, parathyroid hormone, hormone replacement therapy, selective estrogen receptor modulators, calcitonin, calcitriol, glucocorticoids, fluoride, strontium, or anabolic steroids.
25. Have donated > 100 mL blood or plasma within 28 days prior to Randomisation.
26. Have participated in another study with an investigational drug within 60 days prior to Randomisation or are currently participating in or intending to participate in another clinical study of an investigational drug before completion of all scheduled evaluation in this clinical study.
27. Subjects who, in the opinion of the Investigator, are not likely to complete the study for whatever reason.
28. Subject who is the Investigator or any sub-Investigator, research assistant, pharmacist, study coordinator, other staff, or relative thereof directly involved in the conduct of the clinical study.
29. Vulnerable subjects

Ages: 28 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2022-11-09 (Actual)

PRIMARY OUTCOMES:
AUCinf | Day 1 to Day 197
  Area under the concentration-time curve from time zero to infinity
AUClast | Day 1 to Day 197
  Area under the concentration-time curve from time zero to the last quantifiable concentration
Cmax | Day 1 to Day 197
  Maximum serum concentration

SECONDARY OUTCOMES:
Tmax | Day 1 to Day 197
  Time to reach Cmax
Vz/F | Day 1 to Day 197
  Apparent volume of distribution during the terminal phase
λz | Day 1 to Day 197
  Terminal rate constant
t1/2 | Day 1 to Day 197
  Terminal half-life
CL/F | Day 1 to Day 197
  Apparent clearance
%AUCextrap | Day 1 to Day 197
  Percentage of AUCinf due to extrapolation from Tlast to infinity
AUEC for CTX percent inhibition | Day 1 to Day 197
  Area under the effect curve from time zero to Day 197 for serum CTX percent inhibition
Incidence of TEAEs | Day 1 to Day 197
  Experience at least 1 TEAE
Incidence of SAEs | Day 1 to Day 197
  Experience at least 1 SAE
Incidence of ADAs | Day 1 to Day 197
  Incidence of ADAs to denosumab
Incidence of NAbs | Day 1 to Day 197
  Incidence of NAbs to denosumab

CONTACTS AND LOCATIONS:
Overall Officials: Hakim Charfi, MD, Principal Investigator — Biotrial Rennes
Locations (2):
- Biotrial, Newark, New Jersey, United States
- Biotrial Rennes, Rennes, France

REFERENCES:
- [Derived] Lee HA, Kim S, Seo H, Kim S. A phase I, randomized, double-blind, single-dose pharmacokinetic study to evaluate the biosimilarity of SB16 (proposed denosumab biosimilar) with reference denosumab in healthy male subjects. Expert Opin Investig Drugs. 2023 Jul-Dec;32(10):959-966. doi: 10.1080/13543784.2023.2273510. Epub 2023 Nov 6. PMID 37870163